CLINICAL TRIAL: NCT00526318
Title: Trial Protocol for the Treatment of Children With High Risk Neuroblastoma (NB2004-HR)
Brief Title: Combination Chemotherapy Followed by Stem Cell Transplant and Isotretinoin in Treating Young Patients With High-Risk Neuroblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GPOH-NB2004-HR; CDR0000564820 (Registry Identifier: PDQ (Physician Data Query)); UNI-KOELN-161; EU-20661
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Dacarbazine; Doxorubicin; etoposide phosphate; Ifosfamide; Isotretinoin; Melphalan; Topotecan; Vincristine; Vindesine; 3-Iodobenzylguanidine; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide phosphate
Drug: ifosfamide
Drug: isotretinoin
Drug: melphalan
Drug: topotecan hydrochloride
Drug: vincristine sulfate
Drug: vindesine
Procedure: autologous hematopoietic stem cell transplantation
Radiation: iobenguane I 131
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy before an autologous stem cell transplant stops the growth of tumor cells by stopping them from dividing or by killing them. It also prepares the patient's bone marrow for the stem cell transplant. The stem cells are given to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Giving isotretinoin after transplant may kill any remaining tumor cells. It is not yet known which combination chemotherapy regimen is more effective when given before a stem cell transplant and isotretinoin in treating neuroblastoma.

PURPOSE: This randomized clinical trial is studying two different combination chemotherapy regimens to compare how well they work when given before a stem cell transplant and isotretinoin in treating young patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free survival of pediatric patients with high-risk neuroblastoma treated with standard induction chemotherapy vs topotecan hydrochloride-containing induction chemotherapy followed by myeloablative autologous stem cell transplantation and consolidation therapy with isotretinoin.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare early response (complete response, very good partial response, partial response, mixed response, stable disease, and progression/relapse) after 2 courses of standard vs experimental induction chemotherapy (or after 60 days if the second course is not yet finished).
* Compare response to standard vs experimental induction chemotherapy before autologous stem cell transplantation (or after 280 days if induction chemotherapy is not yet finished).
* Compare the toxicity of standard vs experimental induction chemotherapy during courses 1 and 2 and the frequency of ≥ grade 3 toxicity during the last 6 courses of induction chemotherapy.
* Compare the extent of initial surgery and best surgery (biopsy vs incomplete resection vs macroscopic complete resection) and the frequency of complications related to surgery (e.g., nephrectomy, bleeding, infection, or intestinal obstruction).
* Compare the acute and long-term side effects of external-beam radiotherapy.
* Correlate the activity of MIBG and whole-body radiation dose.
* Collect and store tumor material in the tumor bank for future evaluation of other molecular markers (MYCN and status of chromosome 1p and 11q) and prognostic significant gene signatures.

OUTLINE: This is a multicenter study. Patients are stratified according to disease stage, lactate dehydrogenase (LDH) status, MYCN status, and age at diagnosis (stage 4 disease; LDH not elevated; any MYCN status; age at diagnosis 1-21 years vs stage 4 disease; LDH elevated; any MYCN status; age at diagnosis ≥ 1 but < 2 years vs stage 4 disease; LDH elevated; any MYCN status; age at diagnosis 2-21 years vs localized disease; MYCN amplification; age at diagnosis ≥ 6 months)

* Induction chemotherapy: Patients are randomized to 1 of 2 induction chemotherapy arms.

  * Arm I (standard): Patients receive N5 chemotherapy comprising cisplatin IV continuously over 96 hours and etoposide phosphate IV continuously over 96 hours on days 1-4 and vindesine IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 9 and continuing until blood counts recover. Patients then receive N6 chemotherapy comprising vincristine IV over 1 hour on days 1 and 8, dacarbazine IV over 1 hour on days 1-5, ifosfamide IV continuously over 120 hours on days 1-5, and doxorubicin hydrochloride IV over 4 hours on days 6 and 7. Patients also receive G-CSF SC once daily beginning on day 10 and continuing until blood counts recover. Treatment with N5 and N6 chemotherapy alternates every 21 days for 6 courses (N5 chemotherapy is given in courses 1, 3, and 5 and N6 chemotherapy is given in courses 2, 4, and 6).
  * Arm II (experimental): Patients receive N8 chemotherapy comprising cyclophosphamide IV over 1 hour on days 1-7, topotecan hydrochloride IV continuously over 168 hours on days 1-7, and etoposide phosphate IV over 1 hour on days 8-10. Patients also receive G-CSF SC once daily beginning on day 12 and continuing until blood counts recover. Treatment with N8 chemotherapy repeats every 21 days for 2 courses. Patients then receive N5 chemotherapy alternating with N6 chemotherapy as in arm I.
* Surgery: Patients may undergo secondary surgery after completion of 4 or 6 courses of induction chemotherapy but prior to radiotherapy.
* Radiotherapy (131I-MIBG therapy and external-beam radiotherapy [EBRT]): Patients with active residual primary tumor after the completion of induction chemotherapy undergo ^131I-MIBG therapy* prior to autologous stem cell transplantation (ASCT) and EBRT after ASCT.

NOTE: *Patients with MIBG negative neuroblastoma at initial diagnosis will only receive EBRT.

* Myeloablative ASCT: Patients receive melphalan IV over 30 minutes on days -8 to -5, etoposide phosphate IV over 4 hours on day -4, and carboplatin IV over 1 hour on days -4 to -2. Patients undergo reinfusion of CD34+ stem cells on day 0. Patients also receive G-CSF SC or IV over 4 hours once daily beginning on day 2 and continuing until blood counts recover.
* Consolidation therapy (isotretinoin)*: Beginning 30 days after ASCT, patients receive oral isotretinoin once daily on days 1-14. Treatment repeats every 28 days for up to 6 courses. Beginning 3 months later, patients receive an additional 3 courses of isotretinoin.

NOTE: *Isotretinoin must not be given concurrently with radiotherapy

After completion of study treatment, patients are followed every 6 weeks for 1 year, every 3 months for 4 years, and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma according to any of the following criteria:

  * Histological diagnosis from tumor tissue
  * Presence of distinct neuroblastoma cells in the bone marrow and elevated catecholamine metabolites (HVA, VMA) in blood or urine
* High-risk disease, meeting 1 of the following criteria:

  * Stage 4 disease, regardless of the MYCN status (1-21 years of age)
  * Stage 1-3 or 4S disease with MYCN amplification (6 months -21 years of age)

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception (hormonal contraception or intra-uterine device [IUD])

PRIOR CONCURRENT THERAPY:

* No concurrent participation in another clinical trial that would preclude the interventions or outcome assessment of this clinical trial
* No other concurrent anticancer therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2007-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS)

SECONDARY OUTCOMES:
Overall survival (OS)
Impact of well established clinical and molecular risk factors on EFS and OS
Early response, measured after 2 courses of induction chemotherapy
Response to induction therapy, measured before autologous stem cell transplantation
Toxicity during the first 2 courses and the last 6 courses of induction chemotherapy
Impact of the extent of initial and best surgery on outcome and frequency of complications
Acute and late toxicity of radiotherapy
Correlation of MIBG activity with whole-body radiation dose
Molecular markers (MYCN and status of chromosome 1p and 11q)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Berthold, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (68):
- Germany (63):
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Klinikum Bayreuth, Bayreuth
  - Helios Klinikum Berlin, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Evangelisches Krankenhauus Bielfeld, Biefeld
  - Kinderklinik der Universitaet Bonn, Bonn
  - Staedtisches Klinikum - Howedestrase, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Coburg, Coburg
  - Children's Hospital, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Vestische Kinderklinik, Datteln
  - Klinikum Lippe - Detmold, Detmold
  - Klinikum Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Klinikum Duisburg, Duisburg
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Kinderklinik, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitats - Kinderklinik, Greiswald
  - Universitaetsklinikum Halle, Halle
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Gemeinschaftskrankenhaus, Herdecke
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaets - Kinderklinik, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinikum Kemperhof Koblenz, Koblenz
  - Klinikum Krefeld GmbH, Krefeld
  - St. Annastift Krankenhaus, Ludwigshafen
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Staedtisches Klinik - Kinderklinik, Mannheim
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Klinikum Minden, Minden
  - Krankenhaus Muenchen Schwabing, Munich
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Klinikum Neubrandenburg, Neubrandenburg
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Kinderklinik - Universitaetsklinikum Rostock, Rostock
  - Johanniter-Kinderklinik, Sankt Augustin
  - Kinderklink Siegen Deutsches Rotes Kreuz, Siegen
  - Olgahospital, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Universitaets-Kinderspital beider Basel, Basel
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital, Zurich